CLINICAL TRIAL: NCT01887288
Title: Metronomic Capecitabine With Digoxin for Metastatic Breast Cancer Progressing After Anthracycline and Taxane Treatment
Brief Title: Capecitabine With Digoxin for Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Leaving Site
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WRMC 13-05
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Capecitabine with Digoxin (Experimental): Capecitabine PO daily b.i.d., no breaks, starts at day 1 of the first cycle; Digoxin: once daily, starts at day -7 of the first cycle
  (1 cycle - 4 weeks)
  Interventions: Drug: Capecitabine; Drug: Digoxin

INTERVENTIONS:
Drug: Capecitabine — 650 mg/m^2 PO b.i.d.
  Other Names: Xeloda®
Drug: Digoxin — 0.25 mg once daily
  Other Names: Cardoxin®; Digitek®; Lanoxicaps®; Lanoxin®

SUMMARY:
To evaluate the Growth Modulation Index (GMI) of the combination of metronomic capecitabine with oral digoxin in metastatic breast cancer

DETAILED DESCRIPTION:
In this phase II study, the Investigators will combine metronomic capecitabine with digoxin to treat metastatic breast cancer patients who have progressed on both anthracyclines and taxanes. We hypothesize that the combination of digoxin with metronomic capecitabine may lead to increased efficacy and duration of treatment without progression with decreased side effects than standard regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age with histologically confirmed, metastatic breast cancer resistant to anthracyclines and taxanes
2. Anthracycline resistance is defined as tumor progression during treatment or within 3 months of last dose in the metastatic setting, or recurrence within 6 months in the neoadjuvant or adjuvant setting. Alternatively, a minimum cumulative dose of anthracycline of 240 mg/m^2 (doxorubicin) or 360 mg/m^2 (epirubicin) has been reached, or there is contraindication to use anthracycline, the patient is also eligible
3. Taxane resistance is defined as recurrence within 4 months of the last dose in the metastatic setting or within 12 months in the adjuvant setting
4. Having progressed on anti-HER2 or hormonal therapy if they have HER2 positive or hormone-receptor positive breast cancer
5. Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2 and a life expectancy >3 months.
6. Participants must have at least one target lesion as defined by RECIST 1.1 that allows for evaluation of tumor response
7. Absolute neutrophil count ≥ 1500 mm3, platelet count ≥ 100×109 L, hemoglobin ≥ 8.5 g/dL
8. Serum creatinine ≤1.5 times the upper limit of the normal range, total bilirubin ≤ 2 mg/dL, AST/ALT ≤ 5 times the upper limit of normal range
9. No remaining grade 2 or higher toxicity from prior cancer therapies unless judged to be clinically insignificant by the Principal Investigator
10. At least three (3) weeks from prior chemotherapy
11. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must be willing to use an acceptable contraceptive method (abstinence, oral contraceptive or double barrier method) for the duration of the study and for 30 days following the last dose of study drug, and must have a negative urine or serum pregnancy test within 2 weeks prior to beginning treatment on this trial.

Exclusion Criteria:

1. Inadequate renal function with a calculated creatinine clearance less than 51 mL/min.
2. History of ventricular fibrillation, sinus node or AV nodal disease, Wolff Parkinson White Syndrome, hemodynamically significant or life threatening cardiac arrhythmia.
3. Uncontrolled cardiac disease, congestive heart failure, angina or hypertension.
4. Myocardial infarction or unstable angina within 2 months of treatment.
5. Known human immunodeficiency virus (HIV) infection or chronic active Hepatitis B or C (patients are NOT required to be tested for the presence of such viruses prior to therapy on this protocol).
6. Active clinically serious infection > CTCAE (version 4.03) Grade 2.
7. Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
8. Pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 2 within 4 weeks of first dose of study drug.
9. Any other hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks of first dose of study drug.
10. Serious non-healing wound, ulcer, or bone fracture.
11. Major surgery or significant traumatic injury within 2 weeks of first study drug.
12. Inability to complete informed consent process and adhere to the protocol treatment plan and follow-up requirements.
13. Concurrent severe illness such as active infection, or psychiatric illness/social situations that would limit safety and compliance with study requirements.
14. Currently on anti-coagulation therapy with Coumadin, and cannot be switched other forms of anti-coagulation.
15. Patients have symptomatic untreated brain metastasis or leptomeningeal metastases or treated but still symptomatic requiring the use of steroid within the past two weeks.
16. Patients receiving any other investigational agents. Pregnant or Lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiaxin Niu, MD, PhD, Principal Investigator — Western Regional Medical Center
Locations (1):
- Western Regional Medical Center, Goodyear, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Capecitabine With Digoxin: Capecitabine PO daily b.i.d., no breaks, starts at day 1 of the first cycle; Digoxin: once daily, starts at day -7 of the first cycle
  (1 cycle - 4 weeks)
  Capecitabine: 650 mg/m^2 PO b.i.d.
  Digoxin: 0.25 mg once daily
Period: Overall Study
Arm/Group | Capecitabine With Digoxin
Started | 16
Completed | 0
Not Completed | 16
Not completed — The study was terminated and the PI has | 16

BASELINE CHARACTERISTICS:
Population: Data were not collected, The study was terminated due the PI no longer being employed at the site and not having access to the trial information or data.
Arm/Group | Capecitabine With Digoxin
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Metronomic Capecitabine With Oral Digoxin
Description: Evaluate the Growth Modulation Index (GMI) of the combination of metronomic capecitabine with oral digoxin in metastatic breast cancer
Time Frame: One year
Population: data were not collected
Arm/Group | Capecitabine With Digoxin
Number analyzed (Participants) | 0

2. Secondary Outcome: Combination Overall Clinical Benefit by RECIST 1.1
Description: Assess the activity of this combination in terms of overall clinical benefit rates (CBR), including complete response (CR), partial response (PR) or stable disease (SD) as defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Time Frame: One year
Population: data were not collected
Arm/Group | Capecitabine With Digoxin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: data were not collected
Description: data were not collected
Arm/Group | Capecitabine With Digoxin
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes